CLINICAL TRIAL: NCT02948712
Title: Adolescent and Young Adult Survivor Transition (AYAST)
Brief Title: Adolescent and Young Adult Survivor Transition
Acronym: AYAST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE8Z16
Record Dates: First submitted 2016-10-27; First posted 2016-10-28 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Adolescent and Young Adult Cancer
Keywords: distress; survivorship; transition period

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survivor Distress (Experimental): This intervention will use the NCCN Distress Screening Thermometer to score each participant on their level of distress. Depending on the score the intervention will be tailored to the participant based on the Overview of Evaluation and Treatment Schema DIS-4 per the NCCN Distress Guidelines V1.0, 2016.
  Interventions: Behavioral: Distress Screening Thermometer; Behavioral: NCCN Guidelines: Distress management

INTERVENTIONS:
Behavioral: Distress Screening Thermometer — Screening took with an overall distress ranging from 0-10 and additional stress items in the areas of practical problems, family problems, emotional problems, spiritual or religious concerns, and physical problems
Behavioral: NCCN Guidelines: Distress management — Based on the NCCN Guidelines Version 1.0.2016 which recommend brief screening, evaluation, and treatment of distress

SUMMARY:
The purpose of this study is to help adolescents and young adult cancer survivors address their psycho-social needs during the transitional period. The transitional period begins at completion of cancer treatment and continues throughout that first year. Patients often report this period can be difficult and distressing in many areas of life. This study will use a simple tool to measure, on a regular basis, the level of distress a young adult may be feeling. Based on this assessment additional mental health support and intervention can be recommended to help cancer survivors cope and enhance their feelings of well-being.

DETAILED DESCRIPTION:
Study Objective:

To establish a successful distress based intervention program for adolescent and young adult survivors in the transition period.

Study Design and Methods:

The type of design for this study is a feasibility pilot study with repeated measure, within group quantitative design. There is no randomization for this study. The patient will be assessed; at baseline, upon completion of therapy, and at regular three month intervals for the first year, for a total of five assessments. After receiving a referral a member of the AYAST team will contact the patient and set up the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Completed cancer treatment within the past three months of all cancer types and stages
* Signed, written consent

Exclusion Criteria:

* Have not completed cancer treatment within the past three months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Decrease in distress score according to National Comprehensive Cancer Network (NCCN) Guidelines V 1.0.2016 | Up to 15 months after initial visit
  The study coordinators are using the NCCN Distress Screening Thermometer (DST) to screen patients. This includes a using the combined score of the NCCN DST and the associated problem list containing 39 items
  The NCCN Distress Thermometer consists a single-item self- report measure of psychological distress, which consists of an 11-point scale with the endpoints labeled "No distress" (0) and "Extreme distress" (10)

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Baffa, RN, MSN, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States